CLINICAL TRIAL: NCT02852551
Title: A Phase 1, Randomised, Placebo-Controlled, Ascending Single and Multiple Dose Safety, Tolerability, Pharmacokinetic and Food Effect Study of PAT-1251 in Healthy Adult Subjects
Brief Title: Single and Multiple Dose Safety, Tolerability, PK and Food Effect Study of PAT-1251 in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: PharmAkea, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: PAT-1251-CL-001
Record Dates: First submitted 2016-07-15; First posted 2016-08-02 (Estimated); Last update posted 2016-11-30 (Estimated); Status verified 2016-11

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- PAT-1251 Single Dose (Experimental): Oral solution of PAT-1251, 150 - 4000 mg administered once
  Interventions: Drug: PAT-1251
- Placebo Single Dose (Placebo Comparator): Matching placebo solution administered once
  Interventions: Drug: Placebo
- PAT-1251 Multiple Dose (Experimental): Oral tablet(s) of PAT-1251 up to 2000 mg administered daily for 7 days
  Interventions: Drug: PAT-1251
- Placebo Multiple Dose (Experimental): Matching placebo tablets administered daily for 7 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PAT-1251
  Arms: PAT-1251 Multiple Dose; PAT-1251 Single Dose
Drug: Placebo
  Arms: Placebo Multiple Dose; Placebo Single Dose

SUMMARY:
A single-center, randomized, placebo-controlled study consisting of both a single ascending dose (SAD) and a multiple ascending dose (MAD) portion to evaluate the safety, tolerability, pharmacokinetics and effect of food using PAT-1251 orally administered to healthy subjects

ELIGIBILITY:
Inclusion Criteria:

* body mass index (BMI) between 18.0 and 30.0 kg/m2, inclusive
* body weight of 50 to 100 kg, inclusive
* subjects must be in good health

Exclusion Criteria:

* male subjects who do not agree, or whose partners of childbearing potential do not agree, to use appropriate contraception
* female subjects of childbearing potential who do not agree to use 2 acceptable methods of contraception
* history of, any clinically significant major disorder
* clinically significant allergic condition
* significant history of alcoholism or drug/chemical abuse
* use of any tobacco or nicotine-containing products
* clinically significant abnormality in heart rate, blood pressure, temperature, respiration rate, electrocardiogram or clinical laboratory findings
* positive urine drugs of abuse screen or alcohol breath test

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 78 (Actual)
Dates: Start 2016-07; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | one to seven days
  Determination of adverse events will include assessment of vital signs, ECG, clinical laboratory and physical examination

SECONDARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) | one to seven days
Area Under the Plasma Concentration Versus Time Curve (AUC) | one to seven days
Time to Maximum Observed Plasma Concentration (Tmax) | one to seven days
  Comparative pharmacokinetics of single dose administered in a fasted state and following a meal
Terminal elimination half-life (t½) | one to seven days

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Holme, Ph.D., Study Director — PharmAkea, Inc.
Locations (1):
- Covance Clinical Research Unit Ltd., Leeds, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Sponsor Website — http://www.pharmakea.com